CLINICAL TRIAL: NCT06831162
Title: Evaluating the Effectiveness of a Multi-level Health-Related Social Needs Initiative
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Sunil Kripalani, Principal Investigator, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 241778; P50MD017347-03S3 (NIH)
Record Dates: First submitted 2025-02-13; First posted 2025-02-17 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes; Hypertension; Hyperlipidemia; Health-related Social Problems
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multi-level HRSN initiative (Experimental): Eligible patients will receive the HRSN initiative as part of their primary care appointments
  Interventions: Other: Multi-level HRSN initiative

INTERVENTIONS:
Other: Multi-level HRSN initiative — The multi-level health-related social needs (HRSN) initiative includes multiple components aimed at assessing and addressing HRSN in clinical practice: HRSN screening, EHR tools for clinical decision support, training and tools for health care providers to address HRSN, care coordinator support for patient outreach, and community resources for referral and support.

SUMMARY:
The goal of this study is to evaluate the effectiveness of a multi-level health-related social needs (HRSN) initiative among adult patients diagnosed with type 2 diabetes, plus hypertension or hyperlipidemia. The multi-level initiative includes HRSN data collection, training and tools for health care professionals, care coordinator support, and community resources. Patients with type 2 diabetes plus hypertension or hyperlipidemia will be screened for HRSN as part of the primary care clinic intake process to assess if patients have any social needs (like difficulty with getting food, housing, or transportation). If patients screen positive for having social needs, then patients will be offered support, which can include help from primary care providers with adjusting a patient's disease management plan, referrals to care coordinators to provide additional assistance in addressing social needs, and information about community organizations that offer resources for social needs. The initiative will be integrated as a system change across VUMC adult primary care practices.

The investigators will use a prospective, single-arm clinical trial to evaluate effects on clinical outcomes for 12 months. Data will be extracted from the EHR on adult patients diagnosed with type 2 diabetes, and either hypertension or hyperlipidemia. The investigators hypothesize that the initiative will reduce the impact of HRSN on clinical outcomes over the study period. The investigators will also administer surveys to a subgroup of patients to examine trends in self-reported psychosocial and behavioral measures over the course of the initiative.

ELIGIBILITY:
ELIGIBILITY CRITERIA FOR EHR DATA EXTRACTION

Inclusion Criteria:

* 18 years of age or older
* Completed the health-related social needs (HRSN) screener as part of a primary care visit
* Diagnosed with type 2 diabetes, plus hypertension and/or hyperlipidemia as reflected by ICD-10 billing codes
* Receive care at one of six partner Vanderbilt University Medical Center primary care clinics: South One Hundred Oaks, North One Hundred Oaks, Green Hills, Hillsboro Medical Group, Melrose, Bellevue

ELIGIBILITY CRITERIA FOR PATIENT SURVEYS (subset of EHR data)

Inclusion Criteria:

* 18 years of age or older
* Completed the HRSN screener as part of a primary care visit
* Diagnosed with type 2 diabetes
* Receive care at one of six partner Vanderbilt University Medical Center primary care clinics: South One Hundred Oaks, North One Hundred Oaks, Green Hills, Hillsboro Medical Group, Melrose, Bellevue
* English-speaking

Exclusion Criteria:

* Blindness
* Hearing impairment
* Conditions that would interfere with survey completion (e.g., significant dementia, active psychosis or mania)
* Being near the end of life (hospice or home hospice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4809 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-01-24 (Estimated); Study Completion 2026-01-24 (Estimated)

PRIMARY OUTCOMES:
Change in glycemic control | Baseline and 12 months post-baseline
  Hemoglobin A1c extracted from the electronic health record where higher values indicate worse glycemic control.

SECONDARY OUTCOMES:
Change in cholesterol | Baseline and 12 months post-baseline
  Low-density lipoprotein (LDL) extracted from the electronic health record where higher values indicate worse hyperlipidemia.
Change in blood pressure | Baseline and 12 months post-baseline
  Systolic blood pressure extracted from the EHR where higher values indicate worse hypertension.

OTHER OUTCOMES:
Change in medication adherence (survey) | Baseline and 6 months post-baseline
  As assessed by the Adherence to Refills and Medications Scale-Diabetes (ARMS-D) with scores ranging from 11-44, where higher scores indicate more problems with medication adherence (worse).
Change in dietary behavior (survey) | Baseline and 6 months post-baseline
  As assessed by the short version of the Personal Diabetes Questionnaire scale (PDQ-11) Eating Behavior Problems subscale with scores ranging 1-6, where higher scores indicate more problem eating behaviors (worse).
Change in dietary behavior (survey) | Baseline and 6 months post-baseline
  As assessed by the short version of the Personal Diabetes Questionnaire scale (PDQ-11) Use of Information for Decision Making subscale with scores ranging 1-6, where higher scores indicate more use of dietary information for decision making (better).
Change in physical activity (survey) | Baseline and 6 months post-baseline
  As assessed by scores on the Exercise Vital Sign (EVS) Tool with scores ranging 0-1,050 minutes or greater per week of moderate to strenuous physical activity.
Change in diabetes distress (survey) | Baseline and 6 months post-baseline
  As assessed by the Problem Areas in Diabetes-5 (PAID-5) scale with scores ranging from 0 to 20, where higher scores indicate greater diabetes-related emotional distress (worse).
Change in diabetes self-efficacy (survey) | Baseline and 6 months post-baseline
  As assessed by the Perceived Diabetes Self-Management Scale (PDSMS) with scores ranging 8 to 40, where higher scores indicate more self-efficacy (better).
Change in interpersonal processes of care (survey) | Baseline and 6 months post-baseline
  As assessed by the Interpersonal Processes of Care (IPC) survey with scores ranging from 1-5 (calculated as the mean of non-missing responses to the corresponding items), where higher scores indicate higher frequency of the labeled interpersonal process (e.g., decided together; lack of clarity). Scoring occurs for 7 interpersonal processes: lack of clarity; elicited concerns, responded; explained results; decided together; emotional support, compassion; discriminated due to race/ethnicity; and disrespectful office staff.
Change in perceived discrimination (survey) | Baseline and 6 months post-baseline
  As assessed on the Discrimination in Medical Settings scale with scores ranging from 7-35, where higher scores indicate higher frequency of experiences with discrimination in medical settings.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Kripalani, MD, MSc, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
After study results are posted on clinical trials and published, de-identified data will be available upon requests made to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study results are posted on clinical trials and outcomes published in a peer-reviewed journal, until 5 years later
Access Criteria: Contact the principal investigator